CLINICAL TRIAL: NCT05920109
Title: EffecT of eARly analGesia With Erector Spinae Plane Block to Reduce Ventilation After Severe Chest Trauma: a Randomised Control Open-label Trial.
Brief Title: EffecT of eARly analGesia With Erector Spinae Plane Block to Reduce Ventilation After Severe Chest Trauma
Acronym: TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC22.0273
Record Dates: First submitted 2023-05-04; First posted 2023-06-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Severe Chest Trauma
Keywords: chest trauma; erector spinae plane block; Pain management
MeSH Terms: conditions — Thoracic Injuries; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Patients in the experimental group will have a continuous Erector Spinae Plane Block within the first 6 hours post-admission, with a continuous 1ml/h infusion of Ropivacaine (2mg/ml) associated with a 25 ml bolus every 6h.
  Interventions: Procedure: ESP block
- control group (No Intervention): Patients in the control group will receive intravenous multimodal analgesia in the trauma bay. Thoracic epidural analgesia or continuous paravertebral block or serratus plane block will be performed within the first 12 hours post-admission if the pain is not controlled according to our national guidelines.

INTERVENTIONS:
Procedure: ESP block — Patients in the experimental group will have a continuous Erector Spinae Plane Block within the first 6 hours post-admission, with a continuous 1ml/h infusion of Ropivacaine (2mg/ml) associated with a 25 ml bolus every 6h. The catheter will be used from the trauma bay to the ICU as long as possible with a dedicated infusion pump (with a bolus mode). In case of accidental catheter removal, a second introduction of ESP block catheter is allowed within the first 24 hours. In case of continuous ESP block failure (incidence < 5% of the total experimental group), patients will be switched to the control group.
  Arms: experimental group

SUMMARY:
Blunt chest trauma is commonly associated with rib fractures and early pain management is a key goal after chest trauma. In spontaneous breathing patients, pain limits coughing efficiency and secretion clearance, thereby potentially leading to progressive atelectasis, loss of functional residual capacity (FRC) and, ultimately, respiratory distress. In patients under mechanical ventilation, pain interacts with the weaning of mechanical ventilation inducing an increase of the duration of invasive ventilation. According to recent French guidelines for chest trauma management, immediate analgesia is initially performed by intravenous multimodal analgesia followed by a thoracic epidural analgesia or a paravertebral block if the pain is not controlled within the first 12 hours. However, these blocks necessitate an experienced anaesthesiologist, are at risk of severe complications and are contraindicated in case of post-traumatic coagulopathy. All these considerations limit their indication in the trauma bay. The erector spinae plane (ESP) block is an easy to perform, ultrasound guided, regional anaesthesia for pain management after thoracic surgery. This block can be made continuously with a dedicated catheter for a continuous infusion of local anaesthetic drug with boli. The ESP block is performed by depositing the local anaesthetic in the fascial plane, deeper than the erector spinae muscle at the tip of the transverse process of the vertebra. This block is less invasive with fewer contraindications as compared to epidural analgesia or paravertebral blocks. After chest trauma, ESP block was associated with an improvement in respiratory capacity in a retrospective study. However, there is no randomised control trial assessing ESP efficacy. Our hypothesis is that early continuous ESP block in the trauma bay decreases the number of days with invasive and/or non-invasive ventilation after chest trauma.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years

Blunt chest trauma with 3 or more rib fractures on Thoracic CT scan

With spontaneous breathing or under mechanical ventilation in the trauma bay

Requiring an intensive (or intermediate) care unit admission

Exclusion Criteria:

Pre-hospital cardiac arrest

Patient not expected to survive within the first 72 hours

Uncontrolled haemodynamic instability despite initial resuscitation (systolic arterial blood pressure lower than 90 mmHg at the time of catheter insertion)

Mechanical ventilation for severe traumatic brain injury (Abbreviated Injury Score, AIS, head > 2)

Spinal cord injury at the cervical or thoracic levels

Hypovolaemia.

Hypersensitivity to ropivacaine or other amide-bound local anaesthetics

Subject in exclusion period of another interventional study

Pregnant, breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of early analgesia with continuous ESP block after chest trauma on the number of days alive and without invasive or non-invasive ventilation. | 30 days
  The primary endpoint is alive and ventilator free days (VFD) within the first 30 days or hospital discharge, whichever occurred first.

SECONDARY OUTCOMES:
Comparison between the two groups of ESP block feasibility | 48 hours
  Number of failure of catheter placement
Comparison between the two groups of ESP block feasibility | 24 hours
  Time from admission to catheter
Comparison between the two groups of ESP block feasibility | 72 hours
  Number of attempts
Comparison between the two groups of ESP block efficacy | 30 days
  Pain at rest and during physiotherapy and coughing (Numerical Rating Scale : 0 = no pain; 10 = worst possible pain)
Comparison between the two groups of ESP block efficacy | 30 days
  Opioid consumption during ICU stay
Comparison between the two groups of ESP block efficacy | 30 days
  Spirometry parameter (maximum exhaled volume in ml) collected the first seven days of ICU stay (after extubation if mechanically ventilated). The maximal volume collected by the device is 2500 mL.
Comparison between the two groups of ESP block efficacy on chronic pain | 6 months
  Chronic pain assessment with a verbal rating scale (VRS). 0 means no pain, 4 means worst possible pain
Comparison between the two groups of ESP block efficacy on neuropatic pain | 6 months
  neuropathic pain diagnostic questionnaire (DN4). this score can range from 0 to 10 and is positive if greater than or equal to 4/10
Comparison between the two groups of ESP block safety | 48 hours
  Number of haematoma after ESP block puncture
Comparison between the two groups of ESP block safety | 72 hours
  Number of pneumothorax after ESP block catheter insertion
Comparison between the two groups of ESP block safety | 30 days
  Infection of the catheter during ESP block use
Comparison between the two groups of Morbidity and mortality | 30 days
  Number of Hospital Acquired Pneumonia during ICU stay
Comparison between the two groups of Morbidity and mortality | 30 days
  Intubation rate on Day 30
Comparison between the two groups of Morbidity and mortality | 30 days
  ICU-free days within the first 30 days or hospital discharge, whichever occurred first.
Comparison between the two groups of Morbidity and mortality | 30 days
  Mortality at Day one and at Day 30
Comparison between the two groups of Morbidity and mortality | 6 months
  Quality of life at 6 months with EQ-5D-5L questionnaire.
  The EQ-5D-5L descriptive system comprises 5 dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY/DEPRESSION), each dimension has 5 response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the 5 dimensions.
  The EQ VAS records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The EQ VAS provides a quantitative measure of the patient's perception of their overall health.

CONTACTS AND LOCATIONS:
Overall Officials: BOUZAT Pierre, MD, PhD, Principal Investigator — Grenoble Alps University Hospital
Locations (14):
- France (14):
  - CHU Bordeaux - Pellegrin, Bordeaux
  - Hôpital d'instruction des armées Percy, Clamart
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon - AP-HP, Clichy
  - CH Annecy Genevois, Épagny
  - CHU Grenoble Alpes, Grenoble
  - CHU de Lille, Lille
  - Hôpital Pitie Salpetriere - AP-HP, Paris
  - Hôpital Européen Georges Pompidou - AH-HP, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - Hôpital d'Instruction des Armées Sainte Anne, Toulon
  - Chu Toulouse - Hopital Rangueil, Toulouse
  - Chu Toulouse - Hopital Purpan, Toulouse
  - CHRU Hôpitaux De Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veysi VT, Nikolaou VS, Paliobeis C, Efstathopoulos N, Giannoudis PV. Prevalence of chest trauma, associated injuries and mortality: a level I trauma centre experience. Int Orthop. 2009 Oct;33(5):1425-33. doi: 10.1007/s00264-009-0746-9. Epub 2009 Mar 6. PMID 19266199
- [Background] Bachoumas K, Levrat A, Le Thuaut A, Rouleau S, Groyer S, Dupont H, Rooze P, Eisenmann N, Trampont T, Bohe J, Rieu B, Chakarian JC, Godard A, Frederici L, Gelinotte S, Joret A, Roques P, Painvin B, Leroy C, Benedit M, Dopeux L, Soum E, Botoc V, Fartoukh M, Hausermann MH, Kamel T, Morin J, De Varax R, Plantefeve G, Herbland A, Jabaudon M, Duburcq T, Simon C, Chabanne R, Schneider F, Ganster F, Bruel C, Laggoune AS, Bregeaud D, Souweine B, Reignier J, Lascarrou JB. Epidural analgesia in ICU chest trauma patients with fractured ribs: retrospective study of pain control and intubation requirements. Ann Intensive Care. 2020 Aug 27;10(1):116. doi: 10.1186/s13613-020-00733-0. PMID 32852675
- [Background] Huber S, Biberthaler P, Delhey P, Trentzsch H, Winter H, van Griensven M, Lefering R, Huber-Wagner S; Trauma Register DGU. Predictors of poor outcomes after significant chest trauma in multiply injured patients: a retrospective analysis from the German Trauma Registry (Trauma Register DGU(R)). Scand J Trauma Resusc Emerg Med. 2014 Sep 3;22:52. doi: 10.1186/s13049-014-0052-4. PMID 25204466
- [Background] Bouzat P, Raux M, David JS, Tazarourte K, Galinski M, Desmettre T, Garrigue D, Ducros L, Michelet P; Expert's group; Freysz M, Savary D, Rayeh-Pelardy F, Laplace C, Duponq R, Monnin Bares V, D'Journo XB, Boddaert G, Boutonnet M, Pierre S, Leone M, Honnart D, Biais M, Vardon F. Chest trauma: First 48hours management. Anaesth Crit Care Pain Med. 2017 Apr;36(2):135-145. doi: 10.1016/j.accpm.2017.01.003. Epub 2017 Jan 16. PMID 28096063
- [Background] Blondonnet R, Begard M, Jabaudon M, Godet T, Rieu B, Audard J, Lagarde K, Futier E, Pereira B, Bouzat P, Constantin JM. Blunt Chest Trauma and Regional Anesthesia for Analgesia of Multitrauma Patients in French Intensive Care Units: A National Survey. Anesth Analg. 2021 Sep 1;133(3):723-730. doi: 10.1213/ANE.0000000000005442. PMID 33780388
- [Background] Koo CH, Lee HT, Na HS, Ryu JH, Shin HJ. Efficacy of Erector Spinae Plane Block for Analgesia in Thoracic Surgery: A Systematic Review and Meta-Analysis. J Cardiothorac Vasc Anesth. 2022 May;36(5):1387-1395. doi: 10.1053/j.jvca.2021.06.029. Epub 2021 Jun 29. PMID 34301447
- [Background] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545
- [Background] White LD, Riley B, Davis K, Thang C, Mitchell A, Abi-Fares C, Basson W, Anstey C. Safety of Continuous Erector Spinae Catheters in Chest Trauma: A Retrospective Cohort Study. Anesth Analg. 2021 Nov 1;133(5):1296-1302. doi: 10.1213/ANE.0000000000005730. PMID 34473654